CLINICAL TRIAL: NCT06372561
Title: Comparative Evaluation of Melatonin Versus Mineral Trioxide Aggregate on Vital Pulp Therapy in Young Permanent First Molars: An in Vivo Study
Brief Title: Comparative Evaluation of Melatonin Versus MTA on Vital Pulp Therapy in Young Permanent First Molars: An in Vivo Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Melatonin- vital pulp therapy
Record Dates: First submitted 2023-10-31; First posted 2024-04-18 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries in Children; Vital Pulp Therapy
MeSH Terms: interventions — mineral trioxide aggregate; Pemetrexed; Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mineral Trioxide Aggregate (Active Comparator): is a powder that consist of Calcium oxide, silicone dioxide, aluminum oxide, bismuth oxide, purified water. It is a bactericidal dressing material, promotes pulp healing, and does so without producing inflammation and promotes dentin bridge formation.
  Interventions: Drug: Mineral trioxide aggregate (dressing material)
- Melatonin (Experimental): (N-acetyl-5-methoxy-tryptamine) is a pleiotropic hormone synthesized in the pineal gland that has important chronobiotic properties. there is a Melatonin drug (powder) that proved to play an essential role in the regulation of bone growth (bone regeneration) and it may promote osteoblast differentiation, and stimulates mineralized matrix formation
  Interventions: Drug: Melatonin (dressing material)
- Mineral Trioxide and Melatonin (Experimental): Mixture of the two materials' powders.
  Interventions: Drug: Mineral trioxide aggregate (dressing material); Drug: Melatonin (dressing material)

INTERVENTIONS:
Drug: Mineral trioxide aggregate (dressing material) — MTA (Angulus Industrial de productus Odontologists S/a, Brazil) that applied on dental pulp for tissue regeneration
  Other Names: MTA
  Arms: Mineral Trioxide Aggregate; Mineral Trioxide and Melatonin
Drug: Melatonin (dressing material) — melatonin powder 250mg (sigma, Aldrich)- white powder mixing with saline and applied on dental pulp
  Other Names: N-acetyl-5-methoxy-tryptamine
  Arms: Melatonin; Mineral Trioxide and Melatonin

SUMMARY:
The process of dental caries is dynamic and can be either reversible or irreversible depending on the balance between protective and pathologic factors in the oral cavity. Untreated dental caries causes pulpal injury, inflammation, and necrosis. Melatonin plays an essential role in the regulation of bone growth. The actions that melatonin exerts on odontoblasts may be similar to its action on osteoblasts.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and compare the pulp response of young permanent first molars after apexogenesis procedure, using melatonin versus MTA clinically and radiographically. This study will be performed on 45 young permanent first molars that will be divided equally into three groups according to the material used following apexogenesis; GroupI: MTA, GroupII: Melatonin and GroupIII: MTA and Melatonin. apexogenesis procedures will be carried out in children aged 6 to 8 years old. This will be followed by placement of MTA or/and Melatonin material as a sub base in the pulp chamber according to the group. Then, placement of a conventional glass ionomer cement (FUGI IX) as a permanent restoration will be conducted. Then, an immediate postoperative periapical digital x-ray film will be taken for the patients. The patient follow-up will be assigned 1,3,6,9 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1- Apparently healthy and medically free children. 2- Their age ranges from 6-8 years. 3- Both boys and girls will be included. 4- Children should have mandibular permanent first molars with the following clinical and radiographic criteria. 4.1Restorable young permanent first molars. 4.2Absence of clinical evidence of pulp degeneration:
* No history of spontaneous pain, history of night pain or pain that not relieved by analgesics.
* No pain on percussion.
* No mobility.
* Absence of abscess, purulent sinus or soft tissue edema.
* Bleeding should stop within 5 minutes after the amputated pulp stumps.

Exclusion Criteria:

* Internal root resorption.
* External root resorption.
* Inter radicular or periapical bone destruction (radiolucency)
* A deep carious lesion radiologically that approaches the pulp

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-10-02 (Estimated)

PRIMARY OUTCOMES:
Clinically assessment (Modified visual analogue scale) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Pain, sensitivity to percussion (scale values from 0 to 10) 0 means no pain and 10 means the worst pain with failure of the treatment.
Clinically assessment (Millar's index) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  tooth mobility (classes I,II,III) from less mobility to higher mobility.
Clinically assessment (presence or abscence) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  changes in mucobuccal folds (swelling, redness, abscess,fistula)
Radiographic assessment (using Image J software program) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Density of calcific tissue (dentinal bridge) underneath MTA, Melatonin and their mixture (the 3 groups) (Densitometric analysis)
Radiographic assessment (using Image J software program) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Thickness of calcific tissue (dentinal bridge) underneath MTA, Melatonin and their mixture (the 3 groups)
Radiographic assessment (using Image J software program) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Width of apical foramina for the 3 groups.
Radiographic assessment (using Image J software program) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Linear radiographic measurement of root development.
Radiographic assessment (using Image J software program) | Immediately after apexogenesis procedure, after 1 month, 3 months, 6 months, 9 months and 12 months
  Assessment of changes in bone density surrounding the treated teeth (Densiometric analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Gihan GED El-Desouky, Professor, Principal Investigator — Professor; Ghada AH Elbaz, Professor, Principal Investigator — Professor
Locations (1):
- Faculty of Medicine, Suez canal university, Ismailia, Egypt

REFERENCES:
- [Result] Guerrero-Girones J, Alcaina-Lorente A, Ortiz-Ruiz C, Ortiz-Ruiz E, Pecci-Lloret MP, Rodriguez-Lozano FJ, Martinez CM, Ortiz-Ruiz AJ. Melatonin as an Agent for Direct Pulp-Capping Treatment. Int J Environ Res Public Health. 2020 Feb 6;17(3):1043. doi: 10.3390/ijerph17031043. PMID 32041360
- [Result] Liu Q, Fan W, He Y, Zhang F, Guan X, Deng Q, Lu X, He H, Huang F. Effects of melatonin on the proliferation and differentiation of human dental pulp cells. Arch Oral Biol. 2017 Nov;83:33-39. doi: 10.1016/j.archoralbio.2017.06.034. Epub 2017 Jun 30. PMID 28692829
- [Result] Vaseenon S, Chattipakorn N, Chattipakorn SC. Effects of melatonin in wound healing of dental pulp and periodontium: Evidence from in vitro, in vivo and clinical studies. Arch Oral Biol. 2021 Mar;123:105037. doi: 10.1016/j.archoralbio.2020.105037. Epub 2021 Jan 6. PMID 33440268